CLINICAL TRIAL: NCT01875809
Title: Impact of Patient-specific and Procedural Characteristics Like Catecholamine Spill-over on the Long-term Outcome After Renal Denervation and EP Ablation
Brief Title: Impact of Catecholamine Spill-over on Outcome After RDN and EP Ablation
Acronym: RDN-Cath-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Tiroch, Klaus, Privatdozent Dr. med., University of Witten/Herdecke
Other Study IDs: RDN-Cathecholamines-1
Record Dates: First submitted 2013-05-30; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Hypertension
Keywords: RDN; renal denervation; catecholamine; spill-over; blood pressure; electrophysiology; ablation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood for measurement of catecholamines.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Renal denervation (RDN): Change of catecholamine spill-over during RDN
- Electrophysiology (EP) Ablation: Change of catecholamine spill-over during EP ablation

SUMMARY:
Despite a rapidly increasing number of renal denervation (RDN) procedures, only little is known regarding the patient or procedural characteristics influencing the outcome. None of the detectable variables like number of ablation points, temperature rise, impedance drop, have been shown to correlate with the blood pressure (BP) reduction. In this study, the investigators assess different patient and procedural characteristics, like exact patient medication, stress hormones, heart rate variability, and focus on the change of the catecholamine spill-over, and the impact on BP and heart rate after RDN and after EP ablation. The investigators hypothesize the correlation between reduction of catecholamine spill-over due to denervation and the BP reduction. In this study, the investigators will assess 40 patients undergoing RDN and 40 patients undergoing EP ablation.

ELIGIBILITY:
Inclusion Criteria:

* medically-indicated renal denervation
* Age over 18 years
* written informed consent

Exclusion Criteria:

* pregnancy
* expected compliance problems
* current participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing renal denervation or EP Ablation with informed consent fulfilling all inclusion criteria and None of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Catecholamine norepinephrine and epinephrine (pg/ml) | 2 years
  Measurement the differences of norepinephrine and epinephrine (pg/ml) in the renal vein and artery before and after the ablation

SECONDARY OUTCOMES:
Impact of the ablation on 24-hour blood pressure (mmHg) and heart rate (beats/min) | 2 years
  Complete measurement of 24-hour systolic, diastolic, and mean arterial blood pressure (mmHg) and heart rate (beats/min)before and after ablation

CONTACTS AND LOCATIONS:
Overall Officials: Klaus A Tiroch, MD, Principal Investigator — University Wittn/Herdecke
Locations (1):
- HELIOS Klinikum, Wuppertal, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Symplicity HTN-1 Investigators. Catheter-based renal sympathetic denervation for resistant hypertension: durability of blood pressure reduction out to 24 months. Hypertension. 2011 May;57(5):911-7. doi: 10.1161/HYPERTENSIONAHA.110.163014. Epub 2011 Mar 14. PMID 21403086
- [Background] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Result] Schlaich MP, Sobotka PA, Krum H, Lambert E, Esler MD. Renal sympathetic-nerve ablation for uncontrolled hypertension. N Engl J Med. 2009 Aug 27;361(9):932-4. doi: 10.1056/NEJMc0904179. No abstract available. PMID 19710497
- [Derived] Tiroch K, Sause A, Szymanski J, Nover I, Leischik R, Mann JF, Vorpahl M, Seyfarth M. Intraprocedural reduction of the veno-arterial norepinephrine gradient correlates with blood pressure response after renal denervation. EuroIntervention. 2015 Nov;11(7):824-34. doi: 10.4244/EIJV11I7A167. PMID 26603990